CLINICAL TRIAL: NCT02375698
Title: A Phase I, Double-blind, Randomized, Placebo-controlled, Study to Evaluate the Safety and Immunogenicity of AERAS-456 in HIV Negative Adults Successfully Treated for Drug-susceptible Pulmonary Tuberculosis
Brief Title: A Phase I Study of Safety & Immunogenicity of AERAS-456 in HIV-Neg. Adults Treated for Drug-susceptible Pulmonary TB
Acronym: C-037-456
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C-037-456
Record Dates: First submitted 2015-02-20; First posted 2015-03-03 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2017-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gr 1 H56:IC31 5/500 (Experimental): 5ug H56 + 500 ug IC31
  Interventions: Biological: H56:IC31
- Placebo (Placebo Comparator): The placebo consists of 10mM Tris and 169 mM NaCl pH 7.4.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: H56:IC31 — H56:IC31 contains a fusion protein (referred to as H56 antigen, or H56) of 3 mycobacterial antigens (the early secreted antigens Ag85B and ESAT-6, and the latency antigen Rv2660c).
  Other Names: AERAS-456
  Arms: Gr 1 H56:IC31 5/500
Biological: Placebo — The placebo consists of 10mM Tris and 169 mM NaCl pH 7.4.
  Arms: Placebo

SUMMARY:
This is a Phase I, double-blind, randomized, placebo-controlled safety and immunogenicity study in adults who have recently been successfully treated for drug-susceptible pulmonary Tuberculosis (TB). The safety and immunogenicity profile of escalating doses of AERAS-456 in HIV-negative subjects recently treated for drug-susceptible pulmonary TB will be investigated. The study will be conducted at three sites in South Africa.

DETAILED DESCRIPTION:
This study will be the first evaluation of AERAS-456 in subjects who have completed a full course of treatment prescribed for pulmonary TB. Subjects will begin screening for study participation when they have completed 4 calendar months of TB treatment. Subjects meeting the inclusion/exclusion criteria will be randomized within a study group in a 3:1 ratio (N=18 AERAS-456; N=6 placebo) to receive two 0.5 mL intramuscular injections of AERAS-456 or placebo eight weeks apart, on Study Day 0 and Study Day 56.

ELIGIBILITY:
Inclusion Criteria:

1. Is HIV-negative.
2. Is male or female aged 18 through 60 years on Study Day 0.
3. Has completed the written informed consent process.
4. Has a diagnosis of confirmed pulmonary tuberculosis and is on standard TB treatment.
5. Is confirmed to be Mtb negative by either 2 GeneXpert tests or 2 cultures from sputum samples taken on 2 different days at least 1 week apart, the first after at least 4 calendar months of TB treatment and the second day not later than after 5 calendar months (with a window of plus 1 week) of treatment.
6. Agrees to complete the prescribed course of TB treatment (completion of TB treatment can occur after vaccination on Study Day 0; subject must have completed at least 5 calendar months of TB treatment on Study Day 0; if TB treatment is completed before randomization/vaccination then the time from completion of TB treatment to randomization/vaccination should not exceed 28 days).
7. For female subjects: agrees to avoid pregnancy between screening and up until two months after last vaccination. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy from 28 days prior to administration of study vaccine up until two months after the last vaccination. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, or intrauterine device (IUD).
8. Agrees to stay in contact with the study site for the full duration of the study, providing updated contact information as necessary, and has no current plans to move from the study area during the duration of the study.

Exclusion Criteria:

1. Evidence of a new acute illness that may compromise the safety of the subject in the study on Study Day 0.
2. History of TB prior to current episode.
3. TB meningitis or other forms of severe TB with high risk of a poor outcome.
4. Previous medical history that may compromise the safety of the subject in the study, including but not limited to severe impairment of pulmonary function from tuberculosis infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; or uncontrolled epilepsy.
5. Evidence of any systemic disease or any acute or chronic illness that may interfere with the evaluation of the safety of the vaccine.
6. History or laboratory evidence of any possible immunodeficiency state.
7. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
8. Received any non-BCG TB vaccine previously.
9. For female subjects: Currently pregnant, lactating/nursing, or a positive urine HCG.
10. Severe anemia, defined as hemoglobin less than 10 g/dL or a hematocrit less than 30 percent based on screening hematology obtained within 7 days before randomization on Study Day 0.
11. History of autoimmune disease or immunosuppression.
12. Used immunosuppressive medication within 42 days before Study Day 0 (inhaled and topical corticosteroids are permitted).
13. Received immunoglobulin or blood products within 42 days before Study Day 0.
14. Received any investigational drug therapy or investigational vaccine within 6 months before Study Day 0, or planned participation in any other investigational study during the study period.
15. Received any licensed vaccine within 28 days before Study Day 0, or receipt of any vaccine or immunomodulating agent through Study Day 63.
16. Is, in the judgment of the principal investigator, not suitable to participate in this clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dereck Tait, MBChB, Study Director — Aeras
Locations (3):
- South Africa (3):
  - Task Clinical Research Centre, Bellville, Cape Town
  - University of Cape Town Lung Institute, Mowbray, Cape Town
  - The Aurum Institue, Johannesburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tait D, Diacon A, Borges AH, van Brakel E, Hokey D, Rutkowski KT, Hunt DJ, Russell M, Andersen PL, Kromann I, Ruhwald M, Churchyard G, Dawson R. Safety and Immunogenicity of the H56:IC31 Tuberculosis Vaccine Candidate in Adults Successfully Treated for Drug-Susceptible Pulmonary Tuberculosis: A Phase 1 Randomized Trial. J Infect Dis. 2024 Nov 15;230(5):1262-1270. doi: 10.1093/infdis/jiae170. PMID 38557639

RESULTS

PARTICIPANT FLOW:
Groups:
- H56:IC31 5/500: 5ug H56 + 500 ug IC31
  H56:IC31: H56:IC31 contains a fusion protein (referred to as H56 antigen, or H56) of 3 mycobacterial antigens (the early secreted antigens Ag85B and ESAT-6, and the latency antigen Rv2660c).
Period: Overall Study
Arm/Group | H56:IC31 5/500 | Placebo
Started | 16 | 6
Completed | 14 | 4
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H56:IC31 5/500 | Placebo | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 6 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 13 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 0 | 0 | 0
  More than one race | 8 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 16 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Unsolicited AEs: 28 days after each vaccination Solicited AEs: 7 days after each vaccination SAEs: through Day 420 Adverse events of special interest: through Day 420
Time Frame: Day 0 to Day 420
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | H56:IC31 5/500 | Placebo
Number analyzed (Participants) | 16 | 6
Participants
  Participants with any AE | 14 | 6
  Participants with SAEs | 0 | 0

2. Secondary Outcome: Mean Percent Change From Baseline of Participants' Responses to TB Antigens Ag85A and ESAT-6
Description: 13-Color PBMC Intracellular Cytokine Staining (ICS) Assay using PBMCs Percent Antigen-specific T Cell DMSO-subtracted, ANY Cytokine Response - Change from Baseline T Cell: CD4
Time Frame: Day 224
Population: Immunogenicity analysis set
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | H56:IC31 5/500 | Placebo
Number analyzed (Participants) | 14 | 4
Percent change from baseline
  Stimulation Ag: Ag85B | 0.014 (0.0375) | -0.029 (0.0405)
  Stimulation Ag: ESAT-6 | 0.026 (0.0384) | -0.018 (0.0037)

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: for 28 days after each vaccination. Solicited AEs: for 7 days after each vaccination (with diary cards). SAEs: for entire study period (i.e., Study Days 0 to 420). Adverse events of special interest: for entire study period (i.e., Study Days 0 to 420).
Arm/Group | Gr 1 H56:IC31 5/500 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6
Other Adverse Events (participants affected / at risk) | 14/16 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gr 1 H56:IC31 5/500 (N=16) | Placebo (N=6)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 4 (4) | 3 (3)
TACHYCARDIA (Cardiac disorders) | 2 (3) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 4 (5) | 3 (4)
INJECTION SITE ERYTHEMA (General disorders) | 3 (3) | 0 (0)
INJECTION SITE PAIN (General disorders) | 6 (8) | 0 (0)
INJECTION SITE SWELLING (General disorders) | 4 (4) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CONJUNCTIVITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD PRESSURE DIASTOLIC INCREASED (Investigations) | 5 (7) | 0 (0)
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 4 (4) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 3 (4) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (2) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 3 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 3 (4) | 1 (1)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No